CLINICAL TRIAL: NCT05821673
Title: Effect of Argon Plasma Abutment Activation on Soft Tissue Healing: RCT Study With Histological Assessment
Brief Title: Soft Tissue Integration of Different Abutment Surfaces
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Studio Odontoiatrico Associato Dr. P. Cicchese e L. Canullo (Other)
Responsible Party: Principal Investigator, Luigi Canullo, principal investigator; DDS PHD, Studio Odontoiatrico Associato Dr. P. Cicchese e L. Canullo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DD-02
Record Dates: First submitted 2023-04-07; First posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Edentulous Alveolar Ridge; Soft Tissue Healing

STUDY DESIGN:
Intervention Model Description: Participants received either abutments with machine surface characterized by circular micro-threads with a furrow of less than 2 um (surface roughness: Ra=0.2 and Sa=0.11) or abutments with rough Ultrathin Threaded Microsurface with a triangular contour tread with a pitch of 50 μm (surface roughness: Ra=0.62 and Sa=0.60) abutments allocated to the test group were placed in an Argon plasma reactor (Diener Electronic GmbH, Jettingen, Germany) for decontamination and activation. in control group were allocated argon plasma non-treated abutmentsParticipants underwent 2-level randomization for allocation of abutments with different surface configurations and experimental treatment using permuted block technique to limit any selection bias. Allocation concealment was preserved by sealing the tested abutments in sterile envelopes sealed in opaque sleeves opened at the time of the second surgical step.
Who Masked: Participant, Outcomes Assessor
Masking Description: the histologist was blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- abutments with machine surface (Placebo Comparator): abutments with machine surface characterized by circular micro-threads with a furrow of less than 2 um
  Interventions: Procedure: Argon plasma pre-treated abutment insertion; Procedure: abutment insertion
- abutments with rough Ultrathin Threaded Microsurface (Placebo Comparator): abutments with rough Ultrathin Threaded Microsurface with a triangular contour tread with a pitch of 50 μm
  Interventions: Procedure: Argon plasma pre-treated abutment insertion; Procedure: abutment insertion
- argon plasma pre-treated (PT) abutments (Experimental): abutments with rough Ultrathin Threaded Microsurface and abutments with machine surface were pretreated with Argon Plasma
  Interventions: Procedure: Argon plasma pre-treated abutment insertion
- non treated abutments (Placebo Comparator): abutments with rough Ultrathin Threaded Microsurface and abutments with machine surface without Argon Plasma pretreatment.
  Interventions: Procedure: abutment insertion

INTERVENTIONS:
Procedure: Argon plasma pre-treated abutment insertion — abutments allocated to the test group were placed in an Argon plasma reactor (Diener Electronic GmbH, Jettingen, Germany) for decontamination and activation. In order to restrict any post-treatment contamination; abutments were inserted immediately after the end of the plasma process. The reactor was set at 75 W of power and -10 MPa of pressure for 12 min.
  Arms: abutments with machine surface; abutments with rough Ultrathin Threaded Microsurface; argon plasma pre-treated (PT) abutments
Procedure: abutment insertion — the abutments assigned to the control group were screwed onto the implants without receiving argon plasma pretreatment
  Arms: abutments with machine surface; abutments with rough Ultrathin Threaded Microsurface; non treated abutments

SUMMARY:
Objective of the present study was to assess the peri-implant soft tissue profiles between argon plasma pre-treated (PT) and non-treated (NPT) abutments by comparing clinical and histological parameters 2 months after abutment placement.

DETAILED DESCRIPTION:
Patients that need implant supported restoration were recruited for this study. At baseline a specific abutment was screwed at 20 N.Two months following healing abutment placement clinical measurements were evaluated.

Endopoints of the study:

Histological outcomes at 2 using traditional histological staining (ematossilin/eosin) Immunohistological outcomes at 2 using different stainings. Postoperative complications. Comparison between the histological outcomes and the preoperative clinical evaluation of the sites

ELIGIBILITY:
Inclusion Criteria:

1. Patient requiring implant supported restoration.
2. Residual alveolar bone width of edentulous jaw of > 8mm.
3. Keratinized mucosa width of >6mm
4. Males and females between 18-80 years old
5. Patients with healthy periodontal conditions (Treated periodontitis, PI<25%, BoP<25%)
6. Patients that are willing to sign an informed consent and participate in a clinical study
7. Generally fit and healthy and able to undergo oral surgical procedures under local anesthesia.
8. Teeth at the surgical site which required removal were extracted a minimum of 12 weeks prior to sinus floor elevation

Exclusion Criteria:

1. Patients who smoke over 10 cigarettes/day
2. Pregnancy (confirmed by verbal inquiry)
3. Chronic systemic pathologies (e.g. diabetes) and neoplastic of the Oro-Facial District 4.
4. Patients taking bisphosphonates
5. Any sites where an implant already failed sites
6. Untreated Periodontitis
7. Dental sites with acute infections
8. Chronic inflammatory diseases of the oral cavity
9. Autoimmune diseases (cortisone intake)
10. Allergy declared to one or more medicaments to be used during treatment
11. Alcoholics patients and/or drug addicts.
12. History or malignant tumours of the maxillary sinus
13. History of local radiation therapy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2021-12-18 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Histological and immunohistochemical assessment | 2 months after abutment placement
  soft peri-implant tissues and abutment were harvested and histologically processedSpecialized stainings (hematoxylin eosin and picrocirious red) coupled with immunohistochemistry (vimentin, collagen, and CK10) were performed to assess soft tissue inflammation and healing, as well as the collagen content keratinization.
Plaque index (PI) | 2 months after abutment placement
  PI scores were recorded in 6 points around each abutment, averaged, and expressed in %. PI was evaluated with a score of 0,1,2, 3 depending on the amount of plaque at each site.
Bleeding on probing (BoP) | 2 months after abutment placement
  BoP scores were recorded in 6 points around each abutment, averaged, and expressed in %.BoP was used as a dichotomous variable

CONTACTS AND LOCATIONS:
Locations (1):
- Studio Odont.Associato Dr.P.Cicchese E L.Canullo, Rome, Italy/Rome, Italy